CLINICAL TRIAL: NCT07394777
Title: An Open Single-armed Investigation to Evaluate the Safety of pHyph Following a Prolonged Treatment Duration in Adult Women With Bacterial Vaginosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV-2025
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bacterial Vaginosis (BV)
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pHyph treatment (Experimental): 6 doses of pHyph will be administered Day 0-5 and another 6 doses will be administered Day 7-12
  Interventions: Device: pHyph

INTERVENTIONS:
Device: pHyph — pHyph is a vaginal tablet

SUMMARY:
1. Rationale Bacterial vaginosis (BV) is caused by an overgrowth of bacteria and affects most women at some point. The infections can cause foul-smelling discharge and sometimes itching and burning. There are already some approved medications for the treatment of BV. They are not always effective, which means that the infection often returns. Many of these treatments contain antibiotics. In this study, a medical device will be evaluated, a vaginal tablet called pHyph.

   pHyph contains a substance that occurs naturally in the body, Glucono-delta-lactone, which is part of the process when the body handles sugar. It is also an approved food additive. In pHyph, Glucono-delta-lactone restores the acidity of the vagina to normal. In a slightly acidic environment, the bacteria that cause bacterial vaginosis do not thrive, but instead the lactobacilli that are found in a normal vaginal bacterial flora are favored.
2. Aim

Primary aim:

To evaluate the safety after 12 days of treatment with pHyph in patients with BV

Secondary aims:

1. To investigate the difference in the frequency of vaginal dysbiosis after daily treatment for 6 days with pHyph compared to longer daily treatment.
2. To investigate changes in different Lactobacillus species after daily treatment for 6 days with pHyph compared to longer daily treatment.
3. To investigate the difference in clinical efficacy after daily treatment for 6 days with pHyph compared to longer daily treatment.
4. To investigate the relief of the symptom of "fishy odor" after daily treatment for 6 days with pHyph compared to longer daily treatment

Exploratory aims:

To evaluate vaginal microbiome data after different treatment durations in patients with BV 4. Primary outcome measure

To assess the safety and well-tolerated nature of the treatment for patients receiving treatment for a total of 12 days:

1. By monitoring and recording any adverse events that occur during the treatment period, from the first visit to the fourth visit.
2. By assessing for signs of redness, swelling or irritation of the vaginal mucosa using a rating scale from 0 to 3, at days 0, 7, 14 and 25.

5. Secondary outcome measure

The study will compare changes during and after treatment at different time points (days 0, 7, 10, 14 and 25). Among other things, the following are being looked at:

* Presence of bacterial imbalance in the vagina
* Amount of different beneficial Lactobacillus bacteria
* Proportion of patients who recover from symptoms such as foul-smelling or abnormal discharge
* Change in vaginal pH and possible presence of vaginal yeast
* How easy and user-friendly the treatment is perceived according to patients' responses in an app Exploratory outcome measure To further evaluate vaginal microbiome data after different treatment lengths in patients with bacterial vaginosis (BV).

  6. Study design 32 women with BV are planning to be included in the study. The aim is to evaluate the safety after 12 days of treatment (days 0-5 and days 7-12) with pHyph in patients with BV.

  7. Study population The study will include women who have had their period but have not yet reached menopause, are 18 years of age or older and are seeking treatment, directly at a clinic or via advertising, for symptoms of BV, such as foul-smelling or abnormal discharge. The diagnosis of BV is made according to the Amsel criteria, defined as having at least three of the following criteria: thin whitish-yellow discharge, special cells visible under a microscope, a vaginal pH value higher than 4.5, and a distinct fishy odor when a basic substance is added (this symptom must be present). Women with signs of other vaginal infections will not be able to participate in the study.

  8. Interventions The study includes four clinic visits over a period of approximately 25 days. All participants receive active treatment with pHyph vaginal tablets, which are inserted vaginally at home in the evening with a CE marked applicator. Exact instructions are given at the first visit. At the four clinic visits, which are made on days 0, 7, 14 and 25, a gynecological examination is performed and samples are taken. Between visits, participants answer questions about BV symptoms and treatment via a mobile app.
* Visit 1 (Inclusion visit): with information, consent and pregnancy test. A gynecological examination and a sample for BV control are performed. The participant is given an applicator and tablets for 6 days of treatment to use at home every evening.
* Visit 2 (Day 7): A new gynecological examination and a sample for BV control. The participant is given an additional 6 days of tablets. A sample for BV control is taken at home on Day 10.
* Visit 3 (Day 14): A new gynecological examination and a sample for BV control and questions about the ease of use of the product.
* Visit 4 (Day 25): Follow-up visit with a new gynecological examination, sample for BV control, pregnancy test and questions about health and menstruation.

DETAILED DESCRIPTION:
Methodology:

Patients seeking treatment for BV symptoms will be recruited from strategic marketing campaigns, and among possible BV patients managed by clinical sites participating in the investigation.

All patients will receive pHyph treatment for 12 days in total (Day 0-5 + Day 7-12). There will be 4 visits: Visit 1 (Day 0, screening and inclusion), Visit 2 (Day 7), Visit 3 (Day 14), and Visit 4 (Day 25, end-of-investigation). The outcome of the treatment will be compared for the different time points. Microbiome swab samples will be collected at all visits.

At screening (Visit 1), the Investigator or delegated staff will ask patients about the onset and end of their last menstruation. Patients should not be included in the investigation, or inclusion should be postponed, if menstruation is foreseen to occur on Day 0-6 or at the time of Visit 2, scheduled for Day 7. If a patient is menstruating at the scheduled timepoint for Visit 3 or 4, the visit should be re scheduled until the menstrual bleeding is no longer heavy (light bleeding or brown discharge is acceptable), even if this leads to the visit taking place outside the allowed time window.

Patients will self-apply pHyph at home, at night before going to bed, using a vaginal tablet applicator. pHyph and the applicators will be dispensed to the patients at Visit 1 (Day 0) and Visit 2 (Day 7) at the investigation site. To measure pHyph compliance, patients will be asked to return all used and unused pHyph packages, and the number of unused pHyph will be counted.

Patients will continuously complete BV symptom scoring scale questionnaires via the ViedocMe™ mobile application.

Safety assessments:

Local tolerability assessment as well as AE and device deficiency (DD) reporting.

Performance (efficacy) assessments:

Gynaecological exam, including evaluation of Amsel's criteria; vaginal swab for Nugent scoring; vaginal pH assessment; patient questionnaire (BV scoring scale, BV recurrence, usability), vaginal swab for qPCR analysis of vaginal microbiome.

Exploratory assessments:

Additional evaluation of vaginal microbiome DNA data.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the clinical investigation, and to comply with all clinical investigation requirements.
2. Adult, post-menarchal, pre-menopausal women aged 18 years or older.
3. Diagnosis of BV according to Amsel's criteria, defined as having at least 3 of the 4 following criteria:

   * Thin, white, yellow, homogeneous discharge.
   * Clue cells on microscopy (>20% of epithelial cells).
   * pH of vaginal fluid >4.5.
   * Release of "fishy odour", i.e., a positive "whiff test" when alkali (10% KOH solution) is added. This symptom must be present.
4. Negative urine pregnancy test at screening.
5. Willing to refrain from using any intravaginal products (e.g., contraceptive creams, gels, foams, sponges, sex toys, lubricants or tampons, etc.) until Day 14.
6. Willing to use condoms during any sexual intercourse with a male sexual partner until the pHyph treatment is complete (Day 14).
7. Willing to use a method of contraception, e.g., condoms, hormonal contraception (oral, injectable, implantable, intravaginal, or transdermal), IUD (if a copper IUD is used, it must be combined with a condom) or intrauterine hormone-releasing system (IUS), during any sexual intercourse that might result in pregnancy from Visit 1 (Day 0) until Visit 4 (Day 25) to prevent pregnancy.

Exclusion Criteria:

1. Patients with known or apparent signs of other infectious causes of vaginitis (e.g., vulvovaginal candidiasis, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at screening.
2. History of or presence at screening (Day 0) of any other clinically significant disease or disorder, medical/surgical procedure, or trauma, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the clinical investigation, or influence the results or the patient's ability to participate in the clinical investigation.
3. Anticipated menstruation during the first treatment period (Day 0 until Day 7).
4. Patients who are pregnant or breastfeeding.
5. Patients who are planning to conceive within the 25 days of the investigation.
6. Patients who were treated for BV within the 14 days preceding screening.
7. Patients who are currently receiving antibiotic therapy unrelated to BV or have received antibiotic therapy within the 14 days preceding screening.
8. Patients who have used any pH-modifying vaginal products within the 14 days preceding screening.
9. Patients who have received an investigational drug in a clinical trial within 30 days prior to screening.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, to any of the product components.
11. The Investigator considers the patient unlikely to comply with clinical investigation procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety based on reported adverse events from Visit 1 up until the end of Visit 4 and local tolerability based on signs of erythema, oedema and excoriation on the vaginal mucosa, according to a scoring scale (0-3), assessed at each visit. | From enrollment until Day 25

SECONDARY OUTCOMES:
Occurrence of vaginal dysbiosis. | From enrollment until Day 25
  Comparison will be made between the different visits/timepoints
qPCR count of Lactobacillus crispatus | From enrollment until Day 25
  Comparison between the different visits/timepoints
qPCR count of beneficial Lactobacillus species (i.e., all Lactobacillus species except L. iners). | From enrollment until Day 25
qPCR count of all Lactobacillus species | From enrollment until Day 25
Clinical cure rate according to Amsel criteria | From enrollment until Day 25
  Defined as the absence of all of the following 3 Amsel criteria:
  1. Thin, white, yellow, homogenous discharge
  2. Clue cells on microscopy (>20% of epithelial cells)
  3. Release of a "fishy odour", i.e., a positive "whiff test" when alkali (10% potassium hydroxide [KOH] solution) is added.
Proportion of patients that do not have the symptom "fishy odour", as assessed by the Investigator as part of the Amsel criteria. | From enrollment until Day 25
Proportion of patients that do not have the symptom "Thin, white, yellow, homogenous discharge", as assessed by the Investigator as part of the Amsel criteria. | From enrollment until Day 25
Clinical cure rate, defined as Nugent score <4 and defined as Nugent score <7, respectively. | From enrollment until Day 25
  Nugent score is a gram stain scoring system assessing the presence of large Gram-positive rods, small gram-variable rods, and curved gram-variable rods. A score of 7-10 is consistent with bacterial vaginosis (BV), 4-6 is considered intermediate of BV and 0-3 is considered negative for BV
Clinical cure rate, defined as clinical cure according to secondary endpoint 6 (Amsel criteria) and Nugent score <4 or Nugent score <7, respectively, i.e., both criteria have to be fulfilled. | From enrollment until Day 25
  Nugent score is a gram stain scoring system assessing the presence of large Gram-positive rods, small gram-variable rods, and curved gram-variable rods. A score of 7-10 is consistent with bacterial vaginosis (BV), 4-6 is considered intermediate of BV and 0-3 is considered negative for BV.
Proportion of patients that do not have the symptom "fishy odour" after start of treatment, measured by using a patient questionnaire administered via mobile application. | From enrollment until Day 25
Proportion of patients that do not have the symptom "thin abnormal discharge", measured by using a patient questionnaire administered via mobile application. | From enrollment until Day 25
Occurrence of vaginal yeasts, as assessed by analysis of the vaginal microbiome. | From enrollment until Day 25
Vaginal pH | From enrollment until Day 25
Usability measured using a patient questionnaire administered via mobile application on Day 14 | From enrollment until Day 14
  Usability is assessed from dichotomous questions

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - CTC Stockholm, Solna
  - CMedical, Uppsala

IPD SHARING:
Plan to Share IPD: No